CLINICAL TRIAL: NCT00000824
Title: A Pilot Study of HIV Specific Cytotoxic T Lymphocyte (CTL) Therapy in HIV-Infected Patients With CD4+ T Cells 100-350 Cells/mm3
Brief Title: A Study of Cytotoxic T Lymphocyte (CTL) Therapy in HIV-Infected Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: SPIRAT 2
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 1995-04

CONDITIONS: HIV Infections
Keywords: Immunotherapy, Adoptive; T-Lymphocyte Subsets; T-Lymphocytes, Cytotoxic; Dendritic Cells
MeSH Terms: conditions — HIV Infections | interventions — Lymphocyte Count

INTERVENTIONS:
Drug: Lymphocytes, Activated

SUMMARY:
To define the safety of cytotoxic T lymphocytes (CTLs) generated from sibling-supplied dendritic cells and lymphocytes and infused into an HIV-infected patient. To determine the efficacy of these CTLs in helping the immune system to fight HIV.

With lower CD4 counts, HIV-infected patients may not be able to produce dendritic cells and lymphocytes, special types of immune cells that generate HIV-specific CTLs. Infusion of CTLs generated from the dendritic cells and lymphocytes of an HIV-negative sibling may enable the body to recognize HIV more readily and increase immune response against the virus.

DETAILED DESCRIPTION:
With lower CD4 counts, HIV-infected patients may not be able to produce dendritic cells and lymphocytes, special types of immune cells that generate HIV-specific CTLs. Infusion of CTLs generated from the dendritic cells and lymphocytes of an HIV-negative sibling may enable the body to recognize HIV more readily and increase immune response against the virus.

Dendritic cells and lymphocytes are obtained from an HIV-negative sibling. HIV-specific CTLs are generated from these cells and then infused into the HIV-infected patient monthly for 6 months. Siblings must be able to donate on multiple occasions, and patients are followed every 2-4 weeks during the study. Patients are screened over 3 months prior to study entry.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HLA A2+.
* Other HLA matching with sibling.
* CD4 count 100-350 cells/mm3.
* No active opportunistic infection or malignancy (other than cutaneous Kaposi's sarcoma).
* Current stable antiviral regimen.
* Normal lab values and chest x-ray.

Donor siblings must have:

* HLA A2+.
* HIV negativity.
* Good venous access.
* Ability to donate on multiple occasions.
* Negative status for hepatitis B and C.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Immunomodulators.
* Cytokines.
* Systemic steroids.
* IV pentamidine.
* Investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Univ School of Medicine, Stanford, California, United States